CLINICAL TRIAL: NCT01742091
Title: A Multiple Dose Study of LY2541546 to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics in Healthy Postmenopausal Women
Brief Title: A Multiple Dose Study of LY2541546 in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 13405; I2M-MC-GSDE (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: Postmenopausal females; Volunteers
MeSH Terms: interventions — blosozumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 180 mg LY2541546 SC Q4W (Experimental): 180 milligram (mg) LY2541546 administered subcutaneous (SC) once every 4 weeks (Q4W) for 8 weeks. Placebo administered SC at Weeks 2 and 6 to maintain the blind.
  Interventions: Drug: LY2541546 - SC; Drug: Placebo - SC
- 270 mg LY2541546 SC Q2W (Experimental): 270 mg LY2541546 administered (SC) once every 2 weeks (Q2W) for 8 weeks.
  Interventions: Drug: LY2541546 - SC
- 270 mg LY2541546 SC Q4W (Experimental): 270 mg LY2541546 administered (SC) once every 4 weeks (Q4W) for 8 weeks. Placebo administered SC at Weeks 2 and 6 to maintain the blind.
  Interventions: Drug: LY2541546 - SC; Drug: Placebo - SC
- 540 mg LY2541546 IV Q4W (Experimental): 540 mg administered intravenous (IV) once every 4 weeks (Q4W) for 8 weeks. Placebo administered IV at Weeks 2 and 6 to maintain the blind.
  Interventions: Drug: LY2541546 - IV; Drug: Placebo - IV
- 750 mg LY2541546 IV Q2W (Experimental): 750 mg administered (IV) once every 2 weeks (Q2W) for 8 weeks.
  Interventions: Drug: LY2541546 - IV
- Placebo Q2W (Placebo Comparator): Placebo administered IV or SC once every 2 weeks for 8 weeks.
  Interventions: Drug: Placebo - SC; Drug: Placebo - IV

INTERVENTIONS:
Drug: LY2541546 - SC — Administered SC
  Other Names: Blosozumab
  Arms: 180 mg LY2541546 SC Q4W; 270 mg LY2541546 SC Q2W; 270 mg LY2541546 SC Q4W
Drug: LY2541546 - IV — Administered IV
  Other Names: Blosozumab
  Arms: 540 mg LY2541546 IV Q4W; 750 mg LY2541546 IV Q2W
Drug: Placebo - SC — Administered SC
  Arms: 180 mg LY2541546 SC Q4W; 270 mg LY2541546 SC Q4W; Placebo Q2W
Drug: Placebo - IV — Administered IV
  Arms: 540 mg LY2541546 IV Q4W; Placebo Q2W

SUMMARY:
The purpose of this study is to assess the safety and side effects of multiple doses of LY2541546 in postmenopausal women when given subcutaneously (injection just under the skin) and intravenously (directly into a vein). The study will also test how long it takes the study drug to get into the body, how long it takes the body to get rid of it, the overall effect of the study drug on the body, and whether antibodies to the study drug are formed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal females, as determined by medical history and physical examination
* Body mass index (BMI) at screening between 19.0 and 32.0 kilograms per square meter (kg/m^2), inclusive
* Acceptable clinical laboratory test results, blood pressure and heart rate
* Have given written informed consent

Exclusion Criteria:

* Within 30 days of the initial dose of study drug, have received treatment with a drug that has not received regulatory approval for any indication
* Have received study treatment in any trial of an investigational osteoporosis treatment, including LY2561553 (parathyroid hormone receptor modulator), within 12 weeks of screening or 5 half-lives, whichever is longer
* Known allergies to LY2541546, its constituents, or related compounds
* Persons who have previously participated in this study or any other study of LY2541546
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders
* History or presence of low platelet count, bleeding issues or family history of bleeding disorders
* Paget's disease, parathyroid disease, or thyroid disease
* Fracture of a long bone within 12 weeks of screening
* Regular use of known drugs of abuse and/or positive findings on urinary drug screening
* Evidence of human immunodeficiency virus (HIV), hepatitis C, hepatitis B and/or positive for anti-HIV antibodies, hepatitis C antibody, or hepatitis B surface antigen
* Current use of therapies for osteoporosis or use of hormone replacement therapy (HRT) within the previous 12 months
* Blood donation within the last month
* Are unwilling or unable to maintain their normal pattern of alcohol, caffeine, smoking, and exercise from the start to the end of the study or to abide by the clinical research unit restrictions. Note: Average weekly alcohol intake must not exceed 14 units per week
* Are unable or unwilling to refrain from nicotine usage during Clinical Research Unit (CRU) confinement

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 180 mg LY2541546 SC Q4W | 270 mg LY2541546 SC Q2W | 270 mg LY2541546 SC Q4W | 540 mg LY2541546 IV Q4W | 750 mg LY2541546 IV Q2W | Placebo Q2W
Started | 9 | 11 | 10 | 9 | 8 | 12
RECEIVED STUDY DRUG | 9 | 11 | 10 | 9 | 8 | 12
Completed | 9 | 11 | 10 | 8 | 7 | 10
Not Completed | 0 | 0 | 0 | 1 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 180 mg LY2541546 SC Q4W | 270 mg LY2541546 SC Q2W | 270 mg LY2541546 SC Q4W | 540 mg LY2541546 IV Q4W | 750 mg LY2541546 IV Q2W | Placebo Q2W | Total
Number analyzed (Participants) | 9 | 11 | 10 | 9 | 8 | 12 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (5.1) | 57 (5.5) | 56 (7.5) | 57 (8.3) | 66 (8.8) | 62 (10.5) | 59 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 10 | 9 | 8 | 12 | 59
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 4 | 0 | 0 | 4 | 4 | 12
  Black or African American | 0 | 0 | 1 | 1 | 0 | 0 | 2
  White | 9 | 7 | 9 | 8 | 4 | 8 | 45
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 10 | 9 | 8 | 12 | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: An SAE is any AE from this study that results in one of the following outcomes:
  * death
  * initial or prolonged inpatient hospitalization
  * a life-threatening experience (that is, immediate risk of dying)
  * persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * is considered significant by the investigator for any other reason
Time Frame: Day 1 through Day 141
Population: All participants who received study drug.
Measure: Number; unit: participants
Arm/Group | 180 mg LY2541546 SC Q4W | 270 mg LY2541546 SC Q2W | 270 mg LY2541546 SC Q4W | 540 mg LY2541546 IV Q4W | 750 mg LY2541546 IV Q2W | Placebo Q2W
Number analyzed (Participants) | 9 | 11 | 10 | 9 | 8 | 12
participants | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration-Time Curve During Dosing Interval at Steady State (AUCss, 0-tau) of LY2541546
Description: Weekly AUC (AUC[0-tau]) during the first and last dosing interval for each participant receiving LY2541546 is reported.
Time Frame: Day 1 through Day 141
Population: All participants who received study drug and had sufficient evaluable results for PK analysis.
Measure: Mean (Standard Deviation); unit: nanomole x hour per mililiter (nmol*h/mL
Arm/Group | 180 mg LY2541546 SC Q4W | 270 mg LY2541546 SC Q2W | 270 mg LY2541546 SC Q4W | 540 mg LY2541546 IV Q4W | 750 mg LY2541546 IV Q2W
Number analyzed (Participants) | 8 | 11 | 10 | 8 | 7
nanomole x hour per mililiter (nmol*h/mL
  First Dose | 6.77 (2.00) | 18.5 (5.27) | 13.9 (4.73) | 61.2 (7.23) | 167 (11.9)
  Last Dose | 6.85 (2.09) | 38.4 (13.3) | 14.7 (5.45) | 68.9 (11.4) | 332 (54.6)

3. Secondary Outcome: Pharmacodynamics (PD): Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) at Day 85
Description: A BMD test measures the amount of mineral (such as calcium) in a defined area of bone in grams per square centimeter (g/cm²). The least squares (LS) mean was adjusted for baseline lumbar spine BMD and treatment group.
Time Frame: Predose and Day 85
Population: All participants who received study drug and had evaluable BMD results at the analyzed time points.
Measure: Least Squares Mean (90% Confidence Interval); unit: gram per square centimeter (g/cm^2)
Arm/Group | 180 mg LY2541546 SC Q4W | 270 mg LY2541546 SC Q2W | 270 mg LY2541546 SC Q4W | 540 mg LY2541546 IV Q4W | 750 mg LY2541546 IV Q2W | Placebo Q2W
Number analyzed (Participants) | 9 | 11 | 10 | 8 | 7 | 11
gram per square centimeter (g/cm^2) | 0.02 [0.00 to 0.04] | 0.05 [0.03 to 0.06] | 0.03 [0.02 to 0.04] | 0.05 [0.03 to 0.07] | 0.06 [0.04 to 0.08] | 0.00 [-0.01 to 0.02]

4. Secondary Outcome: Immunogenicity: The Number of Participants With Anti-LY2541546 Antibodies
Time Frame: Predose (Day 1) and Postdose (Day 29, 85 and 141)
Population: All participants who received study drug and had evaluable antibody results at the analyzed time points.
Measure: Number; unit: participants
Arm/Group | 180 mg LY2541546 SC Q4W | 270 mg LY2541546 SC Q2W | 270 mg LY2541546 SC Q4W | 540 mg LY2541546 IV Q4W | 750 mg LY2541546 IV Q2W | Placebo Q2W
Number analyzed (Participants) | 9 | 11 | 10 | 9 | 8 | 12
participants
  Day 1 | 0 | 0 | 0 | 0 | 1 | 0
  Day 29 | 1 | 0 | 1 | 0 | 0 | 0
  Day 85 | 3 | 2 | 4 | 0 | 0 | 0
  Day 141 | 3 | 2 | 2 | 1 | 5 | 0

5. Secondary Outcome: Pharmacodynamics (PD): Change From Baseline in N-terminal Propeptide of Procollagen Type 1 (P1NP)
Description: N-terminal propeptide of procollagen type 1 (P1NP) is a main bone formation marker. An increase of P1NP in serum reflects elevated anabolic activities of the bone. Change in P1NP from baseline to post baseline time points was analyzed using the repeated-measures model. Least squares (LS) mean was adjusted for baseline P1NP, treatment group, time (i.e. study day), and interaction between treatment group and time.
Time Frame: Predose, through Day 141
Population: All participants who received study drug and had evaluable P1NP results at the analyzed time points.
Measure: Least Squares Mean (90% Confidence Interval); unit: microgram per liter (ug/L)
Arm/Group | 180 mg LY2541546 SC Q4W | 270 mg LY2541546 SC Q2W | 270 mg LY2541546 SC Q4W | 540 mg LY2541546 IV Q4W | 750 mg LY2541546 IV Q2W | Placebo Q2W
Number analyzed (Participants) | 9 | 11 | 10 | 8 | 7 | 11
microgram per liter (ug/L)
  Day 29 | 20.36 [-4.53 to 45.26] | 121.68 [99.15 to 144.20] | 42.60 [18.98 to 66.23] | 124.47 [98.12 to 150.82] | 134.93 [107.36 to 162.50] | 1.36 [-20.71 to 23.44]
  Day 85 | 1.69 [-15.88 to 19.27] | 24.19 [8.28 to 40.09] | 9.66 [-7.02 to 26.34] | 52.44 [33.72 to 71.16] | 91.06 [71.25 to 110.86] | 4.20 [-11.36 to 19.75]

ADVERSE EVENTS:
Arm/Group | 180 mg LY2541546 SC Q4W | 270 mg LY2541546 SC Q2W | 270 mg LY2541546 SC Q4W | 540 mg LY2541546 IV Q4W | 750 mg LY2541546 IV Q2W | Placebo Q2W
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11 | 0/10 | 0/9 | 1/8 | 0/12
Other Adverse Events (participants affected / at risk) | 7/9 | 11/11 | 7/10 | 5/9 | 7/8 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 180 mg LY2541546 SC Q4W (N=9) | 270 mg LY2541546 SC Q2W (N=11) | 270 mg LY2541546 SC Q4W (N=10) | 540 mg LY2541546 IV Q4W (N=9) | 750 mg LY2541546 IV Q2W (N=8) | Placebo Q2W (N=12)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 180 mg LY2541546 SC Q4W (N=9) | 270 mg LY2541546 SC Q2W (N=11) | 270 mg LY2541546 SC Q4W (N=10) | 540 mg LY2541546 IV Q4W (N=9) | 750 mg LY2541546 IV Q2W (N=8) | Placebo Q2W (N=12)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation Increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival Bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 2 (2)
Chest Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection Site Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection Site Erythema (General disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Haemorrhage (General disorders) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection Site Inflammation (General disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Injection Site Mass (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Injection Site Pain (General disorders) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Injection Site Pruritus (General disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection Site Rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection Site Reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Warmth (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensation of Pressure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel Puncture Site Haematoma (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel Puncture Site Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (3)
Animal Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burns First Degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Thyroid Stimulating Hormone Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head Discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 4 (8) | 1 (1) | 1 (1) | 5 (7)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days